CLINICAL TRIAL: NCT05512260
Title: Towards High, Equal and Informed Participation in Swedish Cancer Screening - the BESTa Project.
Brief Title: Development, Implementation and Evaluation of an Individual Decision Aid in Swedish Cancer Screening Programs
Acronym: BESTa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Karolinska Institutet (Other)
Collaborators: Jonkoping University (Other); Malmö University (Other); Umeå University (Other); Leiden University (Other); Dalarna University (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Kaisa Fritzell, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BESTa
Record Dates: First submitted 2022-06-30; First posted 2022-08-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neoplasm, Colorectal; Neoplasm, Breast; Neoplasm, Ovarian
Keywords: Decision Support Techniques; Shared; Decision Making; Health promotion; Early detection of cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women aged 23 -74 and men aged 60 - 74 invited to population based cancer screening (Other): Women aged 23 -74 targeted for breast cancer, cervical and bowel screening and men aged 60-74 targeted for bowel screening will be invited to the project. Efforts will be made to recruit participants who normally do not participate in research and screening, such as those with various disabilities, participants who live outside society and foreign born.
  Interventions: Device: Individual decision aid (iDA)

INTERVENTIONS:
Device: Individual decision aid (iDA) — A web-based iDA (accessible online with various content), will be developed towards individuals approached to cancer screening, although public and accessible to all who are interested in cancer and screening. DAs in screening usually include information on the disease, screening, screening tests, benefits and harms and some value clarification exercise (e.g., interactive questions) aiming at shedding light on the individual´s values and preferences, knowledge and lifestyle.
  Other Names: Decision aid in paper format

SUMMARY:
Background: Sweden has a long tradition of organized national population-based screening programs. Participation rates differ between programs and regions, are relatively high in some groups, but lower in other. To apply an equity perspective on screening, it is desired that individuals make an informed decision on knowledge rather than ignorance, misconceptions, or fear. Decision Aids (DAs) are set to deliver information about different health care options and to help individuals make visible values connected to the options available. DAs are not meant to guide individuals to choose one option over the another. The advantage of an individual Decision Aid (iDA) is that individuals gain knowledge on cancer and screening entering one webpage with possibility to communicate with health professionals and thereafter make their decision regarding participate. The primary objective is therefore to develop and implement a web-based iDA for individuals invited to cancer screening in Sweden. The secondary objective is to evaluate the implemented web-based iDA.

Methods: This study has an evaluative approach with both a process-, an implementation and an outcome evaluation. Multiple methods will be used including patient reported data, focus group discussions and individual interviews using the think aloud technique. The project is based on the framework from The International Patient Decision Aid Standards (IPDAS) and the proposed model development process for DAs as presented by Coulter et al. Individuals aged 23-74, including women aged (the cervical- and breast- and bowel cancer screening module) and men aged (the bowel cancer screening module), will be included in the developmental process. Efforts will be made to recruit participants with disabilities, who live outside society and who are foreign born.

Discussion: To the best of our knowledge the present study is the first aiming at developing an iDA for usage in Swedish context, The iDA is intended to contribute so that individuals invited to screening base their decision on knowledge and with a clear picture of their values and preferences, rather than ignorance, misconceptions, or fear. Furthermore, the iDA is expected to increase knowledge and raise awareness in general about cancer and cancer screening in society.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE For cancer screening programs to be effective, a high willingness from seemingly healthy individuals to participate is a prerequisite. Participation rates differ and are relatively high in some population groups but at the same time low in other groups. It is well known that individuals with lower socioeconomic status, ethnic minorities and individuals with disabilities participate to a limited extent in cancer screening. A decision aid (DA) is set to deliver information about different health care options and to help individuals make their values visible connected to the options available. Using a DA in connection to cancer screening can increase participation based on knowledge rather than misconception or fear.

The present project is based on the theoretical framework of shared decision making (SDM), with the overarching goal to improve the quality of health care decisions. SDM in this project is based on the work of Charles and Gafni with three cornerstones important for the decision-making process: information/knowledge - to make an informed decision persons need information to gain knowledge about e.g., pros and cons; Values/preferences - persons process their options in relation to attitudes and behaviors; and Involvement - of both the individual and health care professionals.

To date, no DA for any of the screening programs exist in Sweden why this project is warranted. By designing the communication strategies in various ways, regarding information about screening options, and to help individuals construct, clarify and communicate personal values, the researchers intention is to support the decision-making process and to address and acknowledge the equity perspective.

METHODS

Phase 1

Design This study has an evaluative approach encompassing both a process-, an implementation and an outcome evaluation. Multiple methods will be used to answer the research questions including patient reported data, focus group discussions and individual interviews using the think aloud technique. The project is based on the framework from IPDAS and the proposed model development process for DAs, as presented by Coulter et al.

Procedure and outcomes

The procedure will follow the model development process for DAs, applying the following steps:

1. Define scope - a description of breast, cervix and bowel cancer including screening will be formulated, information will be gathered regarding treatment, screening tests, true positive true negative results, risks, and benefits with screening vs. non-screening and detection probabilities. The target audience is all individuals invited to cancer screening.
2. Steering group - a multidisciplinary group will be formed with stakeholders: lay people (aged 23-74), different socioeconomic status and ethnicity, from urban and rural areas, invited to and not invited to screening); clinical experts (oncologists, endoscopists, gastroenterologist, gynecologists, registered nurses, psychologists) and other experts (in psychometry and IT); collaboration partners (The Swedish Association of Local Authorities and Regions - SKR, Regional Cancer Centers - RCC, National Board of Health and Welfare). No disclosed declaration of interest.
3. Design - provision of the iDA in paper format, i.e., a version with the tentative content, including the research and evidence that the iDA is based on as well as a description of the prototype development. The design of the paper version is inspired by the work of Schwartz and colleagues and will be evaluated by lay persons and experts for its content and comprehensibility regarding format (information and descriptions in text and images) and language use.
4. Alpha testing - the web-based iDA will be evaluated for its content, comprehensibility, usability and feasibility, regarding format (information and descriptions in text, spoken animations, images, audio, animated videos, certain clickable words to provide additional information, and interactive questions to help individuals to clarify and express values); language use; setting (web-based) and timing (open for anyone, link will be provided with the invitation).
5. Beta testing - the iDA will be tested in a "real world setting" and evaluated regarding format (information and descriptions in text, spoken animations, images, audio, animated videos, certain clickable words to provide additional information, and interactive questions to help individuals to clarify and express values); language use; setting (web-based) and timing (open for anyone, link will be provided with the invitation).

Data collection During the steps 3-5 data will be collected using different qualitative methods. Data regarding content, format, language use, setting and timing will be generated from focus group discussion and individual interviews. An interview guide with opened-ended questions and optional probe questions will guide the data collection. Participants will be able to choose to participate in a focus group discussion or an individual interview.

During step 3, data regarding the questions, including interactive questions (values and preferences, knowledge, and lifestyle exercises) (step 4) will be generated from concurrent cognitive interviewing where the individual gives a verbal account of their thinking while responding to the interactive questions included in the iDA. The interviews will follow a "think aloud" protocol where individuals are asked to respond to the interactive questions and encouraged to think out loud and to verbalize their thoughts while doing so. This gives an understanding on the perception of each question, as the participants work themselves through the content. In addition, probing questions will be asked when changes in appearance, such as frowning or hesitation occurs and when, or if, the session leader needs further clarification.

Data management Demographic data will be pseudo anonymized, meaning that all personal names will be removed during transcription and all participants in the studies will be given a unique code. A code list will not be established since no personal data is handled. All data will be storage in a secured facility at the Division of Nursing, Karolinska Institutet according to regulations at the university.

Data analyses Data generated from focus group discussions and individual interviews will be analyzed using descriptive and manifest content analysis. Data generated from cognitive interviews applying the "think aloud" method will be compiled and organized according to responses.

Phase 2

Procedure and outcomes After the beta-testing the iDA will be public and accessible for all who are invited and/or interested in the cancer screening programs. To be able to evaluate and develop the iDA further, topics such as digital health literacy, knowledge, values and preferences, decisional conflict, concerns, and risk awareness will be studied with self-reported questions. In addition, demographic questions such as sex, age, educational level, employment will be included as well as questions regarding lifestyle and physical activity. Usability of the iDA including the chat function, helpline, and behavior flow, i.e., how individuals navigate in the iDA will also be scrutinized.

Data collection Data will be collected through self-reported questions included in the iDA.

Data management Questionnaire data will be stored in the web-platform owned by RCC. Extracted data will be pseudo anonymized, meaning that all proper names will be removed during transcription and all participants in the studies will be given a unique code. A code list will not be established since no personal number will be handled. All data will be storage in a secured facility at the Division of Nursing, Karolinska Institutet according to regulations at the university.

Data analyses Data will be analyzed and compared using relevant descriptive and inferential statistics.

First results from the alpha- and beta phases are published, please see reference list.

ELIGIBILITY:
Inclusion Criteria:

* women aged 23 -74
* men aged 60 - 74

Exclusion Criteria:

* none

Ages: 23 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Comprehensibility regarding iDA content | up to 10 months
  The iDA will be evaluated for its content using qualitative methods such as individual interviews, focus group discussions and cognitive interviewing
Usability regarding iDA format | up to 10 months
  The iDA will be evaluated for its usability using qualitative methods such as individual interviews, focus group discussions and cognitive interviewing
Feasibility regarding iDA format | up to 10 months
  The iDA will be evaluated for its feasibility using qualitative methods such as individual interviews, focus group discussions and cognitive interviewing

SECONDARY OUTCOMES:
Self-reported knowledge of cancer and screening | up to 12 months
  Knowledge of cancer and screening of iDA users will be evaluated with self-reported questions including response options such as yes/no/do not know
Self-reported attitudes and preferences to cancer screening | up to 12 months
  Attitudes and preferences to screening of iDA users will be evaluated with self-reported questions including response options such as yes/no/do not know
Self-reported lifestyle behaviors | up to 12 months
  Lifestyle behaviors, such as physical activity, food intake, smoking and alcohol of iDA users will be evaluated with self-reported questions including response options such as yes/no/do not know

OTHER OUTCOMES:
Satisfaction with the iDA and the decision | up to 12 months
  Satisfaction with the iDA and the decision of iDA users will be evaluated with self-reported questions including response options such as yes/no/do not know

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Fritzell, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request

REFERENCES:
- [Background] Schechter MD, Rosecrans JA. D-amphetamine as a discriminative cue: drugs with similar stimulus properties. Eur J Pharmacol. 1973 Feb;21(2):212-6. doi: 10.1016/0014-2999(73)90228-8. No abstract available. PMID 4696103
- [Background] Fritzell K, Hedberg B, Woudstra A, Forsberg A, Sventelius M, Kottorp A, Jervaeus A. Making the BEST decision-the BESTa project development, implementation and evaluation of a digital Decision Aid in Swedish cancer screening programmes- a description of a research project. PLoS One. 2023 Dec 12;18(12):e0294332. doi: 10.1371/journal.pone.0294332. eCollection 2023. PMID 38085710
- [Background] Charles C, Gafni A. The vexing problem of defining the meaning, role and measurement of values in treatment decision-making. J Comp Eff Res. 2014 Mar;3(2):197-209. doi: 10.2217/cer.13.91. PMID 24645693
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Coulter A, Stilwell D, Kryworuchko J, Mullen PD, Ng CJ, van der Weijden T. A systematic development process for patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S2. doi: 10.1186/1472-6947-13-S2-S2. Epub 2013 Nov 29. PMID 24625093
- [Background] Schwartz PH, O'Doherty KC, Bentley C, Schmidt KK, Burgess MM. Layperson Views about the Design and Evaluation of Decision Aids: A Public Deliberation. Med Decis Making. 2021 Jul;41(5):527-539. doi: 10.1177/0272989X21998980. Epub 2021 Apr 5. PMID 33813928
- [Background] Drennan J. Cognitive interviewing: verbal data in the design and pretesting of questionnaires. J Adv Nurs. 2003 Apr;42(1):57-63. doi: 10.1046/j.1365-2648.2003.02579.x. PMID 12641812
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Essink-Bot ML, Dekker E. Equal access to colorectal cancer screening. Lancet. 2016 Feb 20;387(10020):724-6. doi: 10.1016/S0140-6736(15)01221-0. Epub 2015 Dec 9. No abstract available. PMID 26680216
- [Result] Fritzell K, Wangmar J, Hedberg B, Woudstra A, Forsberg A, Kottorp A, Franklin KA, Jervaeus A. Making the BEST Decision-the BESTa Project: Description of the Design and Alpha Phases as Part of the Development of a Digital Decision Aid for Cancer Screening in Sweden. J Cancer Educ. 2025 Apr 26. doi: 10.1007/s13187-025-02633-y. Online ahead of print. PMID 40285812
- See also: The use of think-aloud methods in qualitative research an introduction to think-aloud methods. — http://journals.library.brocku.ca/brocked/index.php/home/article/view/38
- See also: International Patient Decision Aid Standards IPDAS. — http://ipdas.ohri.ca/